CLINICAL TRIAL: NCT02077010
Title: Nebulized Inhaled Milrinone in a Hospitalized Advanced Heart Failure Population
Acronym: iMilrinone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170530
Record Dates: First submitted 2014-02-25; First posted 2014-03-04 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: milrinone; heart failure; cardiomyopathy; inhaled
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inhaled nebulized milrinone (Experimental): Inhaled nebulized milrinone 60mg/4ml every 8 hours using a jet nebulizer
  Interventions: Drug: Inhaled nebulized milrinone

INTERVENTIONS:
Drug: Inhaled nebulized milrinone — inhaled nebulized milrinone 60mg/4ml

SUMMARY:
Patients with end stage heart failure have significant symptoms (including fatigue and shortness of breath) which prevent them from being able to perform most activities of daily living. Milrinone is one of the inotropic medications that has been studied and used in the treatment of end stage heart failure. End stage heart failure patients awaiting a heart transplantation often have to be maintained on IV milrinone 24 hours a day through a chronic IV line. Two problems arise with this therapy. First, the IV line itself creates an opportunity for infection and blood clots, in addition to interfering with patient's quality of life. Second, patients may be exposed to higher levels of milrinone when given IV than are necessary for maintaining their heart's function.

By doing this study the investigators hope to learn if a new way of giving HF patients milrinone can lower the levels of plasma milrinone which may lessen the chance of medication side effects, while still preserving the beneficial effects of milrinone. Additionally if the inhaled route of administration is effective patients may not need to have invasive IV lines to administer the medication (currently standard practice) which can cause other unwanted side effects.

DETAILED DESCRIPTION:
Approximately 5.7 million Americans have heart failure, a leading cause of both morbidity and mortality in the United States. Heart failure was listed as a contributing cause in more than 280,000 deaths in 2008 in the U.S. (1 in 9) and about half of patients diagnosed with heart failure die within 5 years. Patients with end stage heart failure have significant symptoms (including fatigue and dyspnea) which prevent them from being able to perform most activities of daily living. These patients often require repeated or prolonged hospitalizations for disease management which contributes significantly to the cost of heart failure for the United States (34.4 billion each year).

Milrinone, a phosphodiesterase III inhibitor, is one of the inotropic medications that has been studied and used in the treatment of acutely decompensated heart failure. Several studies have evaluated chronic intravenous (IV) inotrope use in end stage heart failure for palliation of symptoms as well as evaluated effect on cost through decreased hospital readmissions. Hauptman et al and Harjai et al demonstrated significant decreases in hospital costs due to reductions in days hospitalized and readmissions after initiation of inotropes including milrinone. However, the concern with IV milrinone use is the possibility of increased mortality associated with therapy despite improved hemodynamics (increased cardiac output, decreased filling pressures) and symptoms as was observed with chronic use of oral inotropes. The OPTIME-CHF study confirmed this concern regarding the use of IV milrinone by reporting increased mortality in patients with New York Heart Association (NYHA) class III-IV ischemic heart failure without hemodynamic compromise as well as statistically significant increases in atrial and ventricular arrhythmias when using intravenous milrinone. For this reason, the American Heart Association/American College of Cardiology practice guidelines, recommend use of IV milrinone only for patients presenting with clinical evidence of hypotension associated with hypo-perfusion and elevated cardiac filling pressures in order to maintain systemic perfusion and preserve end-organ performance. Administration of chronic IV inotropes in heart failure patients with refractory symptoms is categorized as a class IIb indication ("usefulness/efficacy is less well established by expert opinion").

This is a prospective, non-blinded, open-label, phase I clinical trial. We plan to enroll a total of ten patients in two blocks of five. Enrollment will be stopped after the first block of 5 patients to analyze the pharmacokinetics and safety of inhaled milrinone. Patients will have advanced, end-stage HF - and at the discretion of their treating cardiologist who ordered the initial right heart catheterization (RHC) for evaluation of HF therapy, patients will be sent for right heart catheterization (RHC) to determine if inotropic therapy would be beneficial. If the treating cardiologist decides to initiate inotropic therapy based on current guideline-recommended therapies after RHC is performed, the patient will be considered for the trial as long as they meet all inclusion/exclusion criteria.

The investigators goals are two fold:

1. To demonstrate safety by monitoring for pre-specified adverse clinical events and by conducting patient reported questionnaires at 24 and 48 +/- 12 hours.
2. To characterize inhaled milrinone pharmacokinetics. Six plasma samples will be drawn at pre-specified time intervals related to inhaled milrinone delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age > 18 years old
2. Symptomatic Stage D heart failure requiring initiation of inotropic medication at the discretion of their cardiologist
3. Signed informed consent

Exclusion Criteria:

1. Patients incapable of signing informed consent for any reason
2. Patients who are pregnant or breastfeeding
3. Systolic blood pressure less than 85 mmHg prior to randomization
4. Documented allergy or adverse reaction to milrinone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Safety Analysis | A patient questionnaire to ascertain patient reported adverse events will be peformed at 24 hours
  Safety analysis will consist of collecting patient reported adverse events around potential local (respiratory tree) adverse events resulting from the inhalation route and systemic adverse effects resulting from the effects of milrinone itself including ventricular tachycardia (VT), atrial arrhythmias, hypotension, and worsening hypoxia.
Pharmacokinetic analysis | Plasma samples will be drawn around the 4th inhaled dose and after the dose at the following time point of 0.5 hours to assess for serum milirinone concentration fro the trough to be no less than 50ng/ml and the peak to be no greater than 500ng/ml.
  Patient will have serial plasma samples drawn to determine inhaled milrinone pharmacokinetics. A total of six 0.5ml plasma samples will be obtained.
Safety Analysis | A patient questionnaire to ascertain patient reported adverse events will be peformed at 48+/- 12 hours.
  Safety analysis will consist of collecting patient reported adverse events
Pharmacokinetic analysis | Plasma samples will be drawn around the 4th inhaled dose and after the dose at the following time point of 1 hour to assess for serum milirinone concentration fro the trough to be no less than 50ng/ml and the peak to be no greater than 500ng/ml.
  Patient will have serial plasma samples drawn to determine inhaled milrinone pharmacokinetics. A total of six 0.5ml plasma samples will be obtained.
Pharmacokinetic analysis | Plasma samples will be drawn around the 4th inhaled dose and after the dose at the following time point of 2 hours to assess for serum milirinone concentration fro the trough to be no less than 50ng/ml and the peak to be no greater than 500ng/ml.
  Patient will have serial plasma samples drawn to determine inhaled milrinone pharmacokinetics. A total of six 0.5ml plasma samples will be obtained.
Pharmacokinetic analysis | Plasma samples will be drawn around the 4th inhaled dose and after the dose at the following time point of 4 hours to assess for serum milirinone concentration fro the trough to be no less than 50ng/ml and the peak to be no greater than 500ng/ml.
  Patient will have serial plasma samples drawn to determine inhaled milrinone pharmacokinetics. A total of six 0.5ml plasma samples will be obtained.
Pharmacokinetic analysis | Plasma samples will be drawn around the 4th inhaled dose and after the dose at the following time point of 8 hours to assess for serum milirinone concentration fro the trough to be no less than 50ng/ml and the peak to be no greater than 500ng/ml.
  Patient will have serial plasma samples drawn to determine inhaled milrinone pharmacokinetics. A total of six 0.5ml plasma samples will be obtained.

SECONDARY OUTCOMES:
All cause mortality | From date of randomization until study drug is completed (less than or equal to 72 hr after randomization)
  Death from any cause during the study period

OTHER OUTCOMES:
Study Withdrawal Criteria -1 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Hypersensitivity reaction to milrinone: Systemic hypotension (MAP < 60 mmHg for > 30 minutes) plus one of the following: bronchospasm (clinical wheezing) or rash (any type) / urticaria (any type)
Withdrawal criteria - 2 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Acute respiratory failure requiring intubation and mechanical ventilation that is temporally related to inhaled milrinone delivery
Withdrawal criteria - 3 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Deterioration of heart failure by the treating cardiologist's clinical assessment that necessitates additional inotrope/vasopressor support (defined as continuous infusion of dobutamine or dopamine at the time of second right heart catheterization and or assessment of primary outcome)
Withdrawal criteria -4 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Deterioration of heart failure by the treating cardiologists clinical assessment that necessitates additional vasopressor medication support (defined as use of ANY norepinephrine, epinephrine or phenylephrine).
Withdrawal criteria -5 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Deterioration of heart failure by the treating cardiologists clinical assessment that necessitates emergent temporary or durable mechanical circulatory support (ECMO, Impella or LVAD)
Withdrawal criteria -6 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Attending heart failure cardiologist decision at anytime during the study (necessitates discussion with site primary investigator)
Withdrawal criteria -7 | From date of randomization until study drug is completed (less than or equal to 60 hr after randomization)
  Patient choice at anytime during the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Shah, MD, Principal Investigator — University of Kansas; Zachary L Cox, PharmD, Principal Investigator — Vanderbilt University Medical Center/ Lipscomb University College of Pharmacy
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No